CLINICAL TRIAL: NCT02270398
Title: Training Dual-task Balance and Walking in Community-dwelling Older Adults With Chronic Stroke: a Randomized Controlled Trial
Brief Title: Dual-task Training in Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Principal Investigator, Marco Yiu-Chung Pang, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20140714003-01
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Stroke
Keywords: Exercise; Balance; Gait; Community; Rehabilitation; Dual-task
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Pliability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dual-task training group (Experimental): Participants in this group will receive dual-task balance and gait training for half hour and relaxation exercise for another half hour in each session. There will be 3 sessions per week for 8 weeks.
  Interventions: Behavioral: Dual-task training group
- Single-task training group (Active Comparator): This group of subjects will participate in single-task gait and balance activities for half hour and single-task cognitive training in sitting position for another half hour in each session. There will be 3 sessions per week for 8 weeks.
  Interventions: Behavioral: Single-task training group
- Flexibility and strength training group (Active Comparator): The subjects in this group will engage in flexibility exercises and upper limb strengthening exercises for one hour in each session. There will be 3 sessions per week for 8 weeks.
  Interventions: Behavioral: Flexibility and strength training group

INTERVENTIONS:
Behavioral: Dual-task training group — Balance and gait exercises while simultaneously engaging in a secondary cognitive task.
  Arms: Dual-task training group
Behavioral: Single-task training group — Balance/gait exercises and cognitive exercises done separately.
  Arms: Single-task training group
Behavioral: Flexibility and strength training group — Whole-body flexibility exercises, upper limb strengthening exercises.
  Arms: Flexibility and strength training group

SUMMARY:
Background Functional community ambulation not only requires a critical level of postural control and walking skills, but also the ability to engage in cognitive tasks while walking (i.e., dual-task walking) and adapt to the constantly-changing environmental contexts. There is evidence showed that dual-task balance and gait performance is significantly impaired after stroke. Increasing evidence also suggests that dual-task balance and gait performance is useful for predicting falls among individuals with stroke. Considering the high clinical relevance of dual-task balance and gait performance, it is essential that stroke rehabilitation adequately addresses dual-task deficits. Developing specific dual-task balance and gait training to enhance dual-task performance is thus necessary to promote community ambulation and reintegration.

Study Aim The aim of this Introduction Many individuals after stroke continue to cope with residual physical impairments after discharge from hospital. One of the major problems encountered by people after stroke is community reintegration. Functional community ambulation not only requires a critical level of postural control and walking skills, but also the ability to engage in cognitive tasks while walking (i.e., dual-task walking) and adapt to the constantly-changing environmental contexts. There has been an increasing awareness of the importance of dual-task gait performance in community-dwelling individuals with stroke in the past few years.

There is evidence showed that dual-task balance and gait performance is significantly impaired after stroke. Increasing evidence also suggests that dual-task balance and gait performance is useful for predicting falls among individuals with stroke. Considering the high clinical relevance of dual-task balance and gait performance, it is essential that stroke rehabilitation adequately addresses dual-task deficits. Developing specific dual-task balance and gait training to enhance dual-task performance is thus necessary to promote community ambulation and reintegration.

Study Aim This will be a single-blinded randomized controlled trial (RCT).The aim of this study is to examine the efficacy of a dual-task exercise program on cognitive-motor interference in balance and walking tasks, balance self-efficacy, participation in everyday activities, community reintegration and incidence of falls among individuals with chronic stroke.

DETAILED DESCRIPTION:
Introduction Many individuals after stroke continue to cope with residual physical impairments after discharge from hospital. One of the major problems encountered by people after stroke is community reintegration. Functional community ambulation not only requires a critical level of postural control and walking skills, but also the ability to engage in cognitive tasks while walking (i.e., dual-task walking) and adapt to the constantly-changing environmental contexts. There has been an increasing awareness of the importance of dual-task gait performance in community-dwelling individuals with stroke in the past few years.

There is evidence showed that dual-task balance and gait performance is significantly impaired after stroke. Increasing evidence also suggests that dual-task balance and gait performance is useful for predicting falls among individuals with stroke. Considering the high clinical relevance of dual-task balance and gait performance, it is essential that stroke rehabilitation adequately addresses dual-task deficits. Developing specific dual-task balance and gait training to enhance dual-task performance is thus necessary to promote community ambulation and reintegration.

Study Aim The aim of this study is to examine the efficacy of a dual-task exercise program on cognitive-motor interference in balance and walking tasks, balance self-efficacy, participation in everyday activities, community reintegration and incidence of falls among individuals with chronic stroke.

Study design

This will be a single-blinded randomized controlled trial (RCT). After baseline evaluation, subjects will be randomly allocated to one of the three groups: (1) dual-task training group, (2) single-task training group, (3) strengthening and flexibility exercise group (controls), using a 1:1:1 randomization sequence.

Measurements Outcomes will be used to compare the therapeutic effects of the 3 treatment groups. The outcome measurements (except data on incidence of falls) will take place at 3 time points: (1) within one week before initiation of intervention (baseline), (2) within one week after completion of training, (3) 8 weeks after completion of training. The fall data will be collected on a monthly basis until 6 months after termination of the intervention period. All assessments will be performed by a researcher who is blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a stroke
* more than 6 months of stroke onset
* aged 50 years or above
* community-dwelling
* medically stable
* score ≥21 on the Montreal Cognitive Assessment (MoCA)
* score ≤ 25 on the Mini Balance Evaluation Systems Test (Mini-BESTest)
* able to ambulate without physical assistance of another person as determined during the 10-meter walk test
* ability to follow 3-step commands

Exclusion Criteria:

* having neurological conditions other than stroke
* not community-dwelling prior to the stroke event
* significant receptive and expressive aphasia
* severe and uncorrected hearing or visual deficits
* serious musculoskeletal disorders (e.g. amputation)
* serious cardiovascular conditions affecting the ability to participate in exercise training
* pain experienced at rest or movement
* other serious illnesses that preclude participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Timed-up-and-go test with and without dual-task | week 0
  A walking test
Timed-up-and-go test with and without dual-task | week 8
  A walking test
Timed-up-and-go test with and without dual-task | week 16
  A walking test

SECONDARY OUTCOMES:
10-meter walk test with and without dual-task | week 0
  A walking test
10-meter walk test with and without dual-task | week 8
  A walking test
10-meter walk test with and without dual-task | week 16
  A walking test
Sensory organization test with and without dual-task | week 0
  A standing balance test
Sensory organization test with and without dual-task | week 8
  A standing balance test
Sensory organization test with and without dual-task | week 16
  A standing balance test
Obstacle crossing with and without dual-task | week 0
  A walking test
Obstacle crossing with and without dual-task | week 8
  A walking test
Obstacle crossing with and without dual-task | week 16
  A walking test
Mini-Balance Evaluations Systems Test | week 0
  A balance test
Mini-Balance Evaluations Systems Test | week 8
  A balance test
Mini-Balance Evaluations Systems Test | week 16
  A balance test
Activities-specific balance confidence scale | week 0
  A questionnaire
Activities-specific balance confidence scale | week 8
  A questionnaire
Activities-specific balance confidence scale | week 16
  A questionnaire
Stroke Specific Quality of Life Scale | week 0
  A questionnaire
Stroke Specific Quality of Life Scale | week 8
  A questionnaire
Stroke Specific Quality of Life Scale | week 16
  A questionnaire
Motricity Index | week 0
  A muscle strength test
Motricity Index | week 8
  A muscle strength test
Motricity Index | week 16
  A muscle strength test
Chedoke Arm and Hand Activity Inventory | week 0
  An arm function test
Chedoke Arm and Hand Activity Inventory | week 8
  An arm function test
Chedoke Arm and Hand Activity Inventory | week 16
  An arm function test
Frenchay Activities Index | week 0
  A questionnaire
Frenchay Activities Index | week 8
  A questionnaire
Frenchay Activities Index | week 16
  A questionnaire
Tinetti Assessment Tool (Gait) | week 0
  A walking test
Tinetti Assessment Tool (Gait) | week 8
  A walking test
Tinetti Assessment Tool (Gait) | week 16
  A walking test
Incidence of fall | week 0-6 months after training
  fall follow-up using log book and monthly telephone calls
Global Rating of Change score | week 8
  A questionnaire
Global Rating of Change score | week 16
  A questionnaire
Upper limb muscle strength | week 0
  dynamometry test
Upper limb muscle strength | week 8
  dynamometry test
Upper limb muscle strength | week 16
  dynamometry test

CONTACTS AND LOCATIONS:
Overall Officials: Marco YC Pang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Hong Kong Polytechnic University, Hung Hom, Hong Kong

REFERENCES:
- [Background] Said CM, Galea MP, Lythgo N. People with stroke who fail an obstacle crossing task have a higher incidence of falls and utilize different gait patterns compared with people who pass the task. Phys Ther. 2013 Mar;93(3):334-44. doi: 10.2522/ptj.20120200. Epub 2012 Oct 11. PMID 23064734
- [Background] Cockburn J, Haggard P, Cock J, Fordham C. Changing patterns of cognitive-motor interference (CMI) over time during recovery from stroke. Clin Rehabil. 2003 Mar;17(2):167-73. doi: 10.1191/0269215503cr597oa. PMID 12625657
- [Background] Silsupadol P, Lugade V, Shumway-Cook A, van Donkelaar P, Chou LS, Mayr U, Woollacott MH. Training-related changes in dual-task walking performance of elderly persons with balance impairment: a double-blind, randomized controlled trial. Gait Posture. 2009 Jun;29(4):634-9. doi: 10.1016/j.gaitpost.2009.01.006. Epub 2009 Feb 7. PMID 19201610
- [Background] Pichierri G, Wolf P, Murer K, de Bruin ED. Cognitive and cognitive-motor interventions affecting physical functioning: a systematic review. BMC Geriatr. 2011 Jun 8;11:29. doi: 10.1186/1471-2318-11-29. PMID 21651800
- [Background] Yang YR, Wang RY, Chen YC, Kao MJ. Dual-task exercise improves walking ability in chronic stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2007 Oct;88(10):1236-40. doi: 10.1016/j.apmr.2007.06.762. PMID 17908563
- [Derived] Pang MYC, Yang L, Ouyang H, Lam FMH, Huang M, Jehu DA. Dual-Task Exercise Reduces Cognitive-Motor Interference in Walking and Falls After Stroke. Stroke. 2018 Dec;49(12):2990-2998. doi: 10.1161/STROKEAHA.118.022157. PMID 30571419